CLINICAL TRIAL: NCT00843908
Title: A Randomized Study of the Treatment of Urodynamic Stress Incontinence: the Tension Free Vaginal Tape (TVT) Versus the Miniarc Sling.
Brief Title: Tension Free Vaginal Tape (TVT) Versus the Miniarc Sling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Mr Jonathan Duckett, Medway NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07/H1101/112
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Urodynamic Stress Incontinence
Keywords: Stress incontinence; Surgical Treatments; Minislings
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TVT (Active Comparator): Women in this arm will undergo the Tension Free Vaginal Tape procedure
  Interventions: Device: Tension Free Vaginal Tape
- Miniarc (Experimental): Women in this group will undergo the Miniarc suburethral sling procedure
  Interventions: Device: Miniarc

INTERVENTIONS:
Device: Tension Free Vaginal Tape — Tension Free Vaginal Tape inserted in the conventional manner in a theatre environment
  Other Names: Advantage TVT, Boston Scientific
  Arms: TVT
Device: Miniarc — The Miniarc suburethral sling will be inserted in the conventional manner in a theatre environment under general anaesthesia
  Other Names: Miniarc, American Medical Systems
  Arms: Miniarc

SUMMARY:
The aim of this study is to assess whether the Miniarc suburethral sling is equivalent to the TVT in the treatment of women with urodynamic stress incontinence (USI). If equivalence is proven, the advantages to women with USI will be potentially significant since the Miniarc may be carried out as an office based procedure, negating the need for an anaesthetic and hospital admission. The investigators null hypothesis is that there is no difference in subjective or objective outcome between the TVT and the Miniarc in the treatment of USI.

Eligible women will be initially assessed with a full history and examination, King's Health Questionnaire and twin channel subtraction cystometry. They will be randomised (using a series of numbered opaque envelopes) to undergo either the TVT or Miniarc. Follow up will be at 6 weeks, with a subjective outcome measure and at 6 months with a repeat subjective assessment and repeat twin channel cystometry.

DETAILED DESCRIPTION:
Description Randomised, prospective study. Objective and subjective outcomes to be evaluated 6 weeks an d6 months post-operatively.

Study population The number of patients enrolled in the study will be decided after consultation with a statistician.

All patients will be recruited from urogynaecology clinics at Medway Maritime Hospital. They will be female and have a urodynamic diagnosis of stress incontinence, having failed conservative management. Those deemed suitable for the TVT operation will be offered entry to the study.

Randomisation and blinding

Patients who have consented to take part in the study will be randomised to have either a conventional TVT (Group A) or a MiniArc (Group B). Each group will be run in parallel. Method of randomisation - consecutively numbered opaque envelopes detailing type of operation.

Patients will be blinded as to the type of tape used. Due to the obvious differences between the devices, it will not be possible to blind researchers to the type of tape.

Each patient will undergo a pre-operative assessment (which may be incorporated into the initial clinic visit), be admitted as an in-patient for the TVT/Mini-arc procedure, and attend a post-operative assessment visit. This last visit will be the exit point from the study. These are detailed below

Pre-operative Assessment

1. Detailed symptom history and examination
2. 3 day urinary diary
3. King's Quality of Life questionnaire
4. Dual channel normal saline subtracted cystometry at a filling rate of 50-100ml/min whilst supine and standing. 7F double lumen catheter used for all measurements

Surgical Technique

Group A will have the TVT inserted under spinal anaesthesia as described by Ulmsten12. Group B will have the MiniArc tape inserted under spinal anaesthesia. All procedures will be undertaken in an operating theatre environment, and carried out by Mr Duckett or a member of his team who has undergone appropriate training. Patients will be catheterised until 6 hours post-operatively. Those who void with a residual of less than 100mls will be discharged the day after the procedure.

Post-operative assessment

1. Carried out at 6 weeks' post-operatively
2. Symptoms assessed using 3 day urinary diary and Patient Global Impression of Improvement (PGI-I)
3. King's quality of life questionnaire
4. Repeat urodynamic studies as described previously, including voiding cystometry (6 months only)
5. Any complications noted, e.g. readmission to hospital, UTI, voiding difficulties
6. Patient satisfaction will be assessed using a 5 point scale at the follow up visit

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be female
2. Subjective evidence of stress predominant symptoms on symptom specific questionnaire
3. Stress incontinence on urodynamics
4. Patients who are capable of understanding and signing the written consent form for participation in the study
5. Patients must have completed their family
6. Patients must be capable of filling in the symptom diary and micturition diary

Exclusion Criteria:

1. Patients who are medically unfit to undergo surgical intervention.
2. Patients who have undergone previous continence surgery
3. Prolapse beyond the introitus
4. Patients with voiding dysfunction
5. Patients with recurrent urinary tract infections
6. Patients with haematuria of unknown origin or known bladder pathology
7. Patients who are not sure that their family is complete
8. Patients unwilling to use a safe method of contraception following the procedure

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The absence of stress incontinence at 6 weeks ascertained by direct questioning and from the Kings Quality of life questionnaire and the absence at 6 months by the same criteria and by urodynamics. | 6 weeks and 6 months

SECONDARY OUTCOMES:
Quality of life (as measured using the King's Health Questionnaire) | 6 weeks and 6 months
Intra-operative complications, e.g. bladder injury | Time of surgery
Post-operative voiding dysfunction | 0-6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medway Maritime Hospital, Gillingham, Kent, United Kingdom

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839